CLINICAL TRIAL: NCT07389967
Title: Nutrition Awareness Among Women With Non-Metastatic Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 25-2834
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Breast Cancer Metastatic
Keywords: nutrition; diet
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-metastatic breast (Experimental): Women aged 18 or older with a diagnosis of non-metastatic breast cancer and having completed all of their primary treatment for early-stage breast cancer (Stage I, II or II); they can be on endocrine treatment.
  Interventions: Behavioral: Educational Brochure

INTERVENTIONS:
Behavioral: Educational Brochure — The two-page educational brochure is emailed to participants after Questionnaire 2 and before they begin Questionnaire 3.

SUMMARY:
This study explores perspectives of women with non-metastatic breast cancer regarding their willingness and ability to make dietary changes pertaining to foods/food products that may pose a risk to their cancer prognosis and survival.

This is a single-group study conducted entirely online. All study activities, including consent, educational brochure and surveys, will be completed remotely. Participants will receive email invitations to complete questionnaires in REDCap.

Questionnaire 1 will collect sociodemographic information (no PHI) and a brief dietary recall.

Questionnaire 2 will assess identification of ultra-processed foods. Before Questionnaire 3, participants will review a two-page educational flyer explaining the link between diet, obesity, and cancer, with information on unhealthy calories and food processing.

Questionnaire 3 will assess participants' willingness and ability to eat healthier foods and reduce unhealthy foods.

At study completion, participants will receive a thank-you message and a brief satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 -Female
* Diagnosis of non-metastatic breast cancer
* Completion of primary treatment for breast cancer
* No recurrence or metastasis; or no other cancer other than basal or squamous cell
* Willingness to provide a private email address for all study activities
* Ability to read and understand English

Exclusion Criteria:

* Inability to comply with one or more of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Willingness and ability to make dietary changes | Baseline
  the perspectives of women with non-metastatic breast cancer on their willingness and ability to make dietary changes related to specific foods and food products will be assessed. Responses will be collected using a patient-reported questionnaire with a 5-point Likert scale ranging from "Unwilling" to "Very Willing" and "Unable" to "Very Able." Higher scores indicate greater willingness and ability to make healthier dietary choices.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Nyrop, PhD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- UNC Cancer Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials